CLINICAL TRIAL: NCT05463978
Title: A Multi-center Retrospective Chart Review to Evaluate the Safety of Sculptra Aesthetic When Used in Non-facial Areas
Brief Title: Sculptra Chart Review
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 43USSA2110
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: Non-facial Skin Aesthetic Conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Females/Males treated with Sculptra Aesthetic in non-facial areas: Sculptra Aesthetic administration in non-facial areas
  Interventions: Device: Sculptra Aesthetic

INTERVENTIONS:
Device: Sculptra Aesthetic — Sculptra Aesthetic in non-facial areas

SUMMARY:
Multi-center retrospective chart review to evaluate the safety of Sculptra Aesthetic when used in non-facial areas

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been treated at the site with Sculptra Aesthetic in non-facial areas
* Subjects with available information about treatment dates and treatment procedures

Exclusion Criteria:

* Subject that have actively asked not to be involved in a study or registry
* Other conditions that in the Investigator's opinion would exclude the subject from participation ; the condition should be recorded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females/males treated with Sculptra Aesthetic in non-facial areas
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
To evaluate safety of Sculptra Aesthetic when used in non-facial areas | January 2018 to 2022
  AEs related to the product or injection procedure reported in the medical chart

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Galderma Research Site, Pasadena, California
  - Galderma Research Site, San Diego, California
  - Galderma Research Site, Solana Beach, California
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Fort Lauderdale, Florida
  - Site Coordinator, New York, New York
  - Galderma Research Site, New York, New York

IPD SHARING:
Plan to Share IPD: No